CLINICAL TRIAL: NCT06152783
Title: Confocal Laser Microendoscopy (CellTouch) for the Diagnosis of Early Gastric Cancer: A Multicenter Clinical Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Wuxi Hisky Medical Technology Co Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CH-2306
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Early Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A group: The sequence of endoscopy in group A was as follows: white light endoscopy, ME-NBI endoscopy,Confocal laser endomicroscopy.
- B group: The sequence of endoscopy in group B was as follows: white light endoscopy, Confocal laser endomicroscopy, ME-NBI endoscopy.

SUMMARY:
This study is A prospective, randomized, multicenter clinical trial: The study intends to include subjects suspected of early gastric cancer, including 378 subjects with neoplastic lesions and 200 subjects with non-neoplastic lesions. The subjects are divided into two groups by random envelopes, A and B, and the endoscopic diagnosis in different groups is performed in different order (including: White light endoscopy,CellTouch, Magnifying endoscopy with NBI(ME-NBI)). Finally, the gold standard of histopathology was used to evaluate the diagnostic performance of CellTouch in the diagnosis of early gastric cancer.The study hypothesized that the sensitivity and specificity of CellTouch in the diagnosis of early gastric cancer could reach more than 90% and more than 95%.

DETAILED DESCRIPTION:
Objectives:

1. Histopathology was used as the gold standard to evaluate the diagnostic performance of CellTouch in the diagnosis of early gastric cancer.

Secondary Objectives

1. Using histopathology as the gold standard, the diagnostic performance of CellTouch and ME-NBI in the diagnosis of early gastric cancer was compared and analyzed.
2. Histopathology was used as the gold standard to evaluate the diagnostic performance of CellTouch combined with ME-NBI and ME-NBI alone in the diagnosis of early gastric cancer.
3. Histopathology was used as the gold standard to evaluate the diagnostic performance of CellTouch and ME-NBI in the differential diagnosis of low-grade intraepithelial neoplasia and high-grade intraepithelial neoplasia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 70 years;
2. Patients who have recently found suspicious lesions by gastroscopy and need further intensive examination;(Suspicious lesions refer to suspected superficial neoplastic lesions visible under white light endoscopy, including elevation type, flatness type and depression type. According to the Paris classification standard);
3. Patients who willing to provide written informed consent.

Exclusion Criteria:

1. Patients with absolute contraindications to gastroscopy;
2. Patients with advanced gastric cancer;
3. Patients who cannot undergo histopathological examination;
4. Patients who cannot be given general anesthesia;
5. Patients who are pregnant or lactating patients, or prepare to conceive or who are at risk of conception due to lack of effective contraception；
6. Patients with history of drug allergies, such as anesthetics, fluorescein sodium, bowel preparation drugs, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have recently found suspicious lesions by gastroscopy and need further intensive examination;(Suspicious lesions refer to suspected superficial neoplastic lesions visible under white light endoscopy, including elevation type, flatness type and depression type. According to the Paris classification standard).
Sampling Method: Probability Sample
Enrollment: 578 (Estimated)
Dates: Start 2023-11-21 (Estimated); Primary Completion 2024-11-21 (Estimated); Study Completion 2024-11-21 (Estimated)

PRIMARY OUTCOMES:
Histopathology was used as the diagnostic gold standard to evaluate the diagnostic performance of CellTouch in the diagnosis of early gastric cancer. | 30 min
  The diagnostic properties of CellTouch include: sensitivity and specificity.

SECONDARY OUTCOMES:
Using histopathology as the diagnostic gold standard, the diagnostic performance of CellTouch and ME-NBI in early gastric cancer was compared and analyzed. | 30 min
  Diagnostic performance related indexes include: accuracy, sensitivity, specificity, positive predictive value, negative predictive value.
Using histopathology as the diagnostic gold standard, the diagnostic performance of CellTouch combined with ME-NBI and ME-NBI alone in early gastric cancer was compared and analyzed. | 30 min
  Diagnostic performance related indexes include: accuracy, sensitivity, specificity, positive predictive value, negative predictive value.
Using histopathology as the diagnostic gold standard, the diagnostic performance of CellTouch and ME-NBI in the differential diagnosis of low-grade intraepithelial neoplasia and high-grade intraepithelial neoplasia was evaluated. | 30 min
  Diagnostic performance related indexes include: accuracy, sensitivity, specificity, positive predictive value, negative predictive value.

CONTACTS AND LOCATIONS:
Overall Officials: zhen-dong jin, phD, Principal Investigator — Changhai Hospital shanghai
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pilonis ND, Januszewicz W, di Pietro M. Confocal laser endomicroscopy in gastro-intestinal endoscopy: technical aspects and clinical applications. Transl Gastroenterol Hepatol. 2022 Jan 25;7:7. doi: 10.21037/tgh.2020.04.02. eCollection 2022. PMID 35243116
- [Background] Han W, Kong R, Wang N, Bao W, Mao X, Lu J. Confocal Laser Endomicroscopy for Detection of Early Upper Gastrointestinal Cancer. Cancers (Basel). 2023 Jan 26;15(3):776. doi: 10.3390/cancers15030776. PMID 36765734
- [Background] Zhou YW, Zhang LY, Ding SN, Zhang AL, Zhu Y, Chen YX, Zhang QC, Sun LT, Yu JR. Hesitate between confocal laser endomicroscopy and narrow-band imaging: how to choose a better method in the detection of focal precancerous state of gastric cancer. Am J Transl Res. 2022 Jan 15;14(1):55-67. eCollection 2022. PMID 35173829
- [Background] Pang S, Yao H, Jiang C, Zhang Q, Lin R. Confocal Laser Endomicroscopy Can Improve the Diagnosis Rate and Range Assessment of Patients With Conflicting Chronic Atrophic Gastritis Results of White Light Endoscopic and Pathological Diagnosis. Front Oncol. 2022 Mar 24;12:809822. doi: 10.3389/fonc.2022.809822. eCollection 2022. PMID 35402229